CLINICAL TRIAL: NCT03543410
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of SEP-4199 for the Treatment of Major Depressive Episode Associated With Bipolar I Disorder (Bipolar I Depression)
Brief Title: A Clinical Study to Test the Effectiveness of an Investigational Drug to Treat People That Have Major Depressive Episodes When They Have Bipolar 1 Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP380-201; 2018-000103-16 (EudraCT Number)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Depressive Episode; Bipolar 1 Depression
Keywords: Depression, Depressive episode, Bipolar, Bipolar 1, Bipolar 1 depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP-4199 200 mg (Experimental): SEP-4199 200 mg/day (supplied in two 100mg tablets)
  Interventions: Drug: SEP-4199 200 mg
- SEP-4199 400 mg (Experimental): SEP-4199 400 mg/day (supplied in two 200mg tablets)
  Interventions: Drug: SEP-4199 400 mg
- Placebo (Placebo Comparator): Placebo (supplied in two tablets/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-4199 200 mg — SEP-4199 200 mg/day (supplied in two 100mg tablets)
  Arms: SEP-4199 200 mg
Drug: SEP-4199 400 mg — SEP-4199 400 mg/day (supplied in two 200mg tablets
  Arms: SEP-4199 400 mg
Drug: Placebo — Placebo (supplied in two tablets/day)
  Arms: Placebo

SUMMARY:
A clinical study to test the effectiveness of an investigational drug to treat people that have major depressive episodes when they have Bipolar 1 Depression

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, fixed-dose study designed to evaluate the efficacy, safety, and tolerability of treatment with SEP-4199 monotherapy given as 200 mg/day or 400 mg/day compared with placebo for the treatment of major depressive episodes associated with bipolar I disorder (bipolar I depression).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 65 years of age, inclusive, at the time of informed consent with bipolar I disorder, current episode depressed with or without rapid cycling disease course (≥ 4 episodes of mood disturbance but < 8 episodes in the previous 12 months) with or without psychotic features (diagnosed by DSM 5 criteria, and confirmed by the SCID 5 CT). The current episode of major depression associated with bipolar I disorder must be confirmed by the Investigator and noted in the source records.
* Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the investigator.
* Subject or legally acceptable representative must possess an educational level and degree of understanding of English or the local language that enables them to communicate suitably with the Investigator and the study coordinator.
* Subject must have a lifetime history of at least one bipolar manic or mixed manic episode. It is strongly recommended that a reliable informant (e.g., family member or caregiver) be available to confirm this history.
* Subject's current major depressive episode is ≥ 4 weeks and less than 12 months in duration at Screening.
* Subject has a MADRS total score ≥ 22 at both Screening and Baseline.
* Subject has a YMRS total score ≤ 12 at Screening.
* Female subjects of childbearing potential must have a negative serum ß-hCG test at Screening.
* Females who participate in this study must be . one of the following:

  * unable to become pregnant (e.g., postmenopausal, surgically sterile, etc.) -OR-
  * Practicing abstinence or part of an abstinent lifestyle
  * using and willing to continue using a highly effective form of birth control for at least 28 days prior to administration of the first dose of study drug, during the treatment period, and 2 months after completion or premature discontinuation from the study drug.
* Male subjects with partners of child bearing potential must be practicing abstinence, part of an abstinent life style or using protocol-specified methods of birth control. See Section 10.4 for further information on acceptable methods of birth control.
* Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening.
* Subjects with type 2 diabetes are eligible for study inclusion only if all of the following conditions are met within 30 days prior to Screening:

  * Subject's random screening glucose is < 200 mg/dL (11.1 mmol/L).
  * Subject's Hemoglobin A1c (HbA1c) ≤ 7.0%.
  * If a subject is currently being treated with oral anti-diabetic medication(s), the dose must have been stable for at least 30 days prior to screening. Such medication may be adjusted or discontinued during the study, as clinically indicated.
  * Subject has not required hospitalization for diabetes or related complications in the past 12 months.
  * Note: Subjects with type 2 diabetes that is newly diagnosed during screening are ineligible for the study.
* Subject who requires concomitant medication treatment with the following agents may be included if they have been on stable doses for the specified times: 1) oral hypoglycemics must be stabilized for at least 30 days prior to baseline; 2) thyroid hormone replacement must be stable for at least 90 days prior to baseline; 3) anti hypertensive agents must be stable for at least 30 days prior to baseline. The subject's medical condition should be deemed clinically stable following consultation with the Medical Monitor as needed.

Exclusion Criteria:

* Subject has a lifelong history or presence of symptoms consistent with a major psychiatric disorder other than bipolar I disorder as defined by DSM 5. Exclusionary disorders include but are not limited to moderate to severe alcohol use disorder (within past 12 months), substance use disorder (other than nicotine or caffeine) within past 12 months, bipolar II disorder, schizoaffective disorder, obsessive compulsive disorder, posttraumatic stress disorder.
* Subject demonstrates a decrease (improvement) of ≥ 25% in MADRS total score from Screening to Baseline, or subject's MADRS total score is < 22 at Baseline.
* Subject has received treatment with antidepressants within 3 days of randomization, fluoxetine at any time within 28 days, an MAO inhibitor within 21 days or clozapine within 120 days. All other psychotropic medications with the exceptions of lorazepam, temazepam,eszopiclone, zopiclone, zolpidem and zolpidem CR require 3 days minimum washout. Depot neuroleptics must be discontinued at least one treatment cycle prior to randomization.
* Subject has suspected/confirmed Borderline Personality Disorder
* Subject currently has a clinically significant neurological, metabolic (including type 1 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorder such as unstable angina, congestive heart failure (uncontrolled), or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study. Subjects with a known history of HIV seropositivity will be excluded.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if under control) must be discussed with the Medical Monitor before being randomized in the study.

* Subject has evidence of any chronic organic disease of the CNS such as tumors, inflammation, active (or history of) seizure disorder, vascular disorder, Parkinson's disease, Alzheimer's disease or other forms of dementia, myasthenia gravis, or other degenerative processes. In addition, subjects must not have a history of intellectual disability or persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, is not exclusionary.
* Subject has a history of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Subjects with pituitary tumors of any duration are excluded.
* Subject demonstrates evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation (use screening values for laboratory evaluation). Subject has a history of stomach or intestinal surgery or any other condition that could interfere with absorption, distribution, metabolism, or excretion of medications.
* Subject has knowledge of any kind of cardiovascular disorder/condition known to increase the possibility of QT prolongation or history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome or Brugada Syndrome) or cardiac conduction disorders, or requires treatment with an antiarrhythmic medication.
* Subject has family history of QTc prolongation or of unexplainable sudden death at < 50 years of age.
* Abnormal 12 lead ECG at Screening, including:

  * QTcF > 450 ms (male subjects) or > 470 ms (female subjects)
  * QRS > 110 ms
  * PR > 200 ms
  * Second- or third-degree atrioventricular block
  * Any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant
* Subject has a history of neuroleptic malignant syndrome (NMS).
* Subject exhibits evidence of severe tardive dyskinesia, severe dystonia, or any other severe movement disorder. Severity is to be determined by the investigator.
* Subject has been diagnosed with type 1 diabetes, or insulin-dependent diabetics.
* Subject who has any abnormal laboratory parameter at screening that indicates a clinically significant medical condition as determined by the investigator. Subjects with fasting blood glucose at screening ≥ 126 mg/dL (7.0 mmol/L) will be excluded from the study. Subjects with fasting blood glucose from 100-125 mg/dL (5.6-6.9 mmol/L) may enter the study based on the approval of the Medical Monitor. Subjects with HbA1c > 7.0% will be excluded. Subjects who are found to have been non-fasting at Screening may be allowed if their blood glucose is < 200 mg/dL. Subjects with random (nonfasting) blood glucose at screening ≥ 200 mg/dL (11.1 mmol/L) must be retested in a fasted state. Subjects with HbA1c > 7.0% will be excluded.
* Subject has a prolactin concentration > 100 ng/mL at screening or have a history of pituitary adenoma.
* Subject has a body mass index (BMI) ≥ 40 or < 18 kg/m2.
* Subject has a history of non-response to an adequate (6-week) trial of three or more antidepressants (with or without mood stabilizers) during the current episode.
* Subject is considered by the Investigator to be at imminent risk of suicide or injury to self, others, or answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at the Screening visit (in the past month [30 days]) or Baseline.
* Subject tests positive for drugs of abuse at screening or baseline. In the event a subject tests positive for cannabinoids (tetrahydrocannabinol), the investigator will evaluate the subject's ability to abstain from cannabis during the study. This information will be discussed with the Medical Monitor for study enrollment consideration.
* Subject has a history of hypersensitivity to more than two distinct chemical classes of drug (e.g., sulfas and penicillins).
* Subjects have received depot neuroleptics unless the last injection was at least one treatment cycle before randomization.
* Subject requires treatment with a drug that consistently prolongs the QTc interval
* Subject has received ECT within 90 days prior to randomization or is expected to require ECT during the study course.
* Subject is currently participating, or has participated in a study with an investigational or marketed compound or device within 6 months prior to signing the informed consent, or has participated in 3 or more studies within 18 months prior to signing the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (87):
- United States (7):
  - CNS Research Science, Inc., Cerritos, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Artemis Insitute for Clinical Research, San Diego, California
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Eastside Therapeutic Resource dba Core Clinical Research, Everett, Washington
- Bulgaria (6):
  - Mental Health Centre -Prof. Dr. Ivan Temkov - Burgas EOOD, Burgas
  - State Psychiatric Hospital-Kardzhali, Kardzhali
  - MHAT-Dr. Hristo Stambolski EOOD, Department of Psychiatry, Kazanlak
  - Mental Health Center - Ruse EOOD, Rousse
  - Neli Nikolova Todorova, MD ,State Psychatric Hospital - s. Tsarev brod, Shumen
  - Mental Health Center - Sofia EOOD, Sofia
- Japan (35):
  - Fukuoka University Hospital, Fukuoka
  - Hatakeyama Clinic, Department of Psychiatry, Fukuoka
  - Hiro Mental Clinic, Department of Psychiatry, Fukuoka
  - Kokura Mental Clinic, Fukuoka
  - Kuramitsu Hospital, Department of Psychiatry, Fukuoka
  - Shinseikai Kaku Mental Clinic, Department of Psychiatry, Fukuoka
  - Someikai Kanagami Clinic, Department of Psychiatry, Fukuoka
  - Jisenkai Nanko Psychiatric Institute, Department of Psychiatry, Fukushima
  - Takahashi Psychiatric Clinic, Hyōgo
  - Azamino Mental clinic, Department of Psychiatry, Kanagawa
  - Medical Corporation Seishinkai Kishiro Mental Clinic, Department of Psychiatry, Kanagawa
  - Musashikosugi J. Kokorono Clinic, Kanagawa
  - Yokohama Onoecho Clinic, Department of Psychiatry, Kanagawa
  - Yutaka Clinic, Kanagawa
  - SagaArashiyama / Tanaka Clinic, Department of Psychiatry, Kyoto
  - Minami-aoyama Anique Street Clinic, Department of Psychiatry, Minato-Ku, Tokyo
  - Clinic Sophia, Okayama
  - Nagaokai Neyagawa Sanitorium, Osaka
  - Asakayama Hospital, Osaka
  - Koshokai Ainhanazono Hospital, Osaka
  - Osaka Institute of Clinical Psychiatry Shin-abuyama Hospital, Osaka
  - Etoh Mental Clinic Meguro, Department of Psychiatry, Tokyo
  - Himorogi Psychiatric Institute, Department of Psychiatry, Tokyo
  - JCHO Yokyo Shinjuku Medical Center, Tokyo
  - Jisenkai Hozumi Himorogi Clinic, Department of Psychiatry, Tokyo
  - Maynds Tower Mental Clinic, Department of Psychiatry, Tokyo
  - Nishi-shinjuku Concieria Clnic, Tokyo
  - Ohwa Mental clinic, Department of Psychiatry, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Department of Psychiatry, Tokyo
  - Sangenjaya Neurology-Psychosomatic Clinic, Department of Psychiatry, Tokyo
  - Senzoku Psychosomatic Clinic, Department of Psychiatry, Tokyo
  - Shinjuku Research Park Clinic, Tokyo
  - Tamaki Clinic, Department of Psychiatry, Tokyo
  - Uguisudani Mental Clinic, Department of Psychiatry, Tokyo
  - Yoyogi Mental Clinic, Tokyo
- Poland (7):
  - Przychodnia Srodmiescie Sp. z.o.o., Bydgoszcz
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Specjalistyczna Praktyka Lekarska Marek Domanski, Lublin
  - Filip Rybakowski Specjalistyczna Praktka Lekarska, Poznan
  - Poradnia Zdrowia Psychicznego "Syntonia", Pruszcz Gdański
  - Gabinet Lekarski Torunskie Centrum PsychiatriI NEUROMED, Torun
  - Osrodek Badan Klinicznych Clinsante Spolka Cywilna, Torun
- Russia (10):
  - Lipetsk regional psychoneurological hospital, Lipetsk
  - State Budgetary Institution of Healthare of the City of Moscow "Psychiatric clinical Hospital #4 n.a. P.B. Gannushkin of the Department of Healthcare of the City o Moscow" Branch "Psychiatric hospital n.a. V.A. Gilyarovsky", Moscow
  - State Budgetary Institution of Healthcare of Nizhniy Novgorod region "Clinical Psychiatric Hospital #1 of Nizhniy Novgorod", Nizhny Novgorod
  - Budgetary Institution of Healthcare of Omsk region "Clinical Psychiatric Hospital named after N.N. Solodnikov", Omsk
  - Limited Liability Company "Treatment and Rehabilitational Scientific Center Phoenix", Rostov-on-Don
  - Saint Petersburg State Institution of Healthcare "Psychiatric Hospital of Sain Nikolai hudotvorets ", Saint Petersburg
  - Federal State Budgetary Institution "National Medical Research Centre of psychiatry and nuerology named after V.M. Bekhterev" of the Ministry of Healthcare of the Russian Federation, department #12, Saint Petersburg
  - Stain Petersburg State Budgetary Institution of Healthcare "Psychoneurological Dispensary #1", Saint Petersburg
  - State Institution of Healtcare "Regional Clinical Psychiatric Hospital of Saint Sofia", Saratov
  - Limited Liability Company "Clinic StoLet", Tomsk
- Serbia (7):
  - Bel Medic General Hospital, Belgrade
  - Clinical Center "Dr. Dragisa Misovic-Dedinje", Belgrade
  - Clinical Center of Serbia, Belgrade
  - General Hospital Euromedik, Belgrade
  - Institute of Mental Health, Belgrade
  - Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - Clinical Center Kragujevac, Kragujevac
- Slovakia (5):
  - Vavrusova Consulting s.r.o. Psychiatricka ambulancia, Bratislava
  - Investa spol. s.r.o., Kosice Psychiatricka ambulancia, Košice
  - Psycholine s.r.0. Psychiatricka ambulancia, Rimavská Sobota
  - Centrum zdravia R.B.K. Psychiatricka ambulancia, Svidník
  - Crystal Comfort s.r.o. Psychiatricka ambulancia, Vranov nad Topľou
- Ukraine (10):
  - Regional Psychoneurological Hospital #3, Department of Neurosis and Borderline States # 8, Ivano-Frankivsk
  - State Institution Institue of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Unit of Emergency sychiatry and Narcology, Kharkiv
  - State Institution Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Unit of Borderline Psychiatry, Kharkiv
  - CI Kherson Regional Psychiatric Hospital of Kherson Regional Council, Male Dep of Psychiatry #3, Female Dep of Psychiatry #10, Kherson
  - Communal Institution (CI) of Kyiv Regional Council regional Psychiatric and Narcological Medical Assocation, Dep #10 (male), Dep #2 (female), Kyiv
  - Communal Institution Odesa regional Medical Center of Mental Health, Dep #6 (Male), Dep #12 (Female), Odesa
  - Communal Institution Odesa Regional Psychiatric Hospital #2, Department #14 (female), Department #16 (male), Odesa
  - Communal Institution Cherkasy regional Psychiatric Hospital of Cherkasy Regional Council, Female Department #11, Male Department #12, Smila
  - Transcarpathian Regional Narcological Dispensary, Department of Psychiatry, Uzhhorod
  - communal Institution Acad. O.I. Yushchenko Vinnytsia Regional Psychoneurological hosital, Male Deparmtent #14, Female Department #15, Vinnytsia M.I. Pyrogov National Medical University, Chair of Psychiatry, Narcology and Psychotherapy with the Course of P, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study may be made available upon request via the Vivli Center for Global Clinical Research Data website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available upon request within 12 months of posting the study results on ct.gov.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://vivli.org

REFERENCES:
- [Derived] Hopkins SC, Tomioka S, Szabo ST, Koblan KS. A clinical trial inclusion criteria to enrich for patients presenting with canonical symptom structure in bipolar depression. Contemp Clin Trials. 2024 Oct;145:107644. doi: 10.1016/j.cct.2024.107644. Epub 2024 Aug 3. PMID 39098761
- [Derived] Hopkins SC, Wilkinson S, Corriveau TJ, Nishikawa H, Nakamichi K, Loebel A, Koblan KS. Discovery of Nonracemic Amisulpride to Maximize Benefit/Risk of 5-HT7 and D2 Receptor Antagonism for the Treatment of Mood Disorders. Clin Pharmacol Ther. 2021 Sep;110(3):808-815. doi: 10.1002/cpt.2282. Epub 2021 Jun 12. PMID 33961287

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 344 subjects were randomized in this study. Three subjects, who were randomized but never received any dose of study medication, were not included in the reporting.
Period: Overall Study
Arm/Group | SEP-4199 200 mg | SEP-4199 400 mg | Placebo
Started | 113 | 114 | 114
Completed | 92 | 101 | 99
Not Completed | 21 | 13 | 15
Not completed — Adverse Event | 10 | 8 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 8
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Due to COVID-19 | 4 | 0 | 2
Not completed — NON-COMPLIANCE WITH STUDY DRUG | 0 | 0 | 2
Not completed — Not Due to COVID-19 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SEP-4199 200 mg | SEP-4199 400 mg | Placebo | Total
Number analyzed (Participants) | 113 | 114 | 114 | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 1 | 3
  Between 18 and 65 years | 112 | 111 | 113 | 336
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (11.65) | 44.4 (12.72) | 43.3 (12.10) | 43.2 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 76 | 64 | 209
  Male | 44 | 38 | 50 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 110 | 109 | 112 | 331
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 16 | 16 | 17 | 49
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 1 | 4
  Black or African American | 6 | 8 | 8 | 22
  White | 89 | 87 | 88 | 264
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Europe | 83 | 82 | 84 | 249
  Japan | 16 | 16 | 17 | 49
  United States | 14 | 16 | 13 | 43
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 113 | 112 | 114 | 339
  >=65 years | 0 | 2 | 0 | 2
Country Name [Count of Participants; unit: Participants]
  Bulgaria | 11 | 10 | 22 | 43
  Japan | 16 | 16 | 17 | 49
  Poland | 5 | 1 | 5 | 11
  Russia | 18 | 20 | 8 | 46
  Serbia | 19 | 26 | 18 | 63
  Slovakia | 8 | 5 | 6 | 19
  Ukraine | 22 | 20 | 25 | 67
  United States | 14 | 16 | 13 | 43
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 75.3 (14.47) | 74.8 (16.19) | 77.5 (16.59) | 75.9 (15.78)
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4.53) | 26.6 (4.91) | 27 (4.94) | 26.6 (4.79)
Baseline BMI Category [Count of Participants; unit: Participants]
  < 18.5 kg/m^2 | 0 | 3 | 0 | 3
  18.5 - <25.0 kg/m^2 | 51 | 50 | 45 | 146
  25.0 - <30.0 kg/m^2 | 42 | 33 | 40 | 115
  >=30.0 kg/m^2 | 20 | 28 | 29 | 77
Baseline Montgomery-Asberg Depression Rating Scale( MADRS )Total Score [Mean (Standard Deviation); unit: units on a scale] — MADRS is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts, each ranging from 0 to 6. The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
  units on a scale | 33.5 (5.77) | 33.8 (5.63) | 34.1 (5.35) | 33.8 (5.58)
Baseline global severity assessed by the Clinical Global Impressions -Severity Depression Score [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions - Severity: Bipolar Version (CGI-BP-S) score (depression) is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
  units on a scale | 4.8 (0.66) | 4.8 (0.65) | 4.9 (0.70) | 4.8 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: MADRS is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts, each ranging from 0 to 6. The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
Time Frame: 6 Weeks
Population: ITT population, excluding subjects from Japan Region
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-4199 200 mg | SEP-4199 400 mg | Placebo
Number analyzed (Participants) | 96 | 97 | 96
units on a scale | -19.485 (1.226) | -19.324 (1.182) | -16.196 (1.231)
Statistical Analysis 1: Comparison: SEP-4199 200 mg vs Placebo; Test type: Superiority; p = 0.044, Mixed Models Analysis — nominal p-value; Mean Difference (Final Values) = -3.290, 95% CI 2-sided [-6.489 to -0.090], Standard Error of Mean 1.625
Statistical Analysis 2: Comparison: SEP-4199 400 mg vs Placebo; Test type: Superiority; p = 0.051, Mixed Models Analysis — nominal p-value; Mean Difference (Final Values) = -3.128, 95% CI 2-sided [-6.273 to 0.017], Standard Error of Mean 1.597

2. Secondary Outcome: Change From Baseline in Global Severity Assessed by the Clinical Global Impressions - Severity: Bipolar Version (CGI-BP-S) Score (Depression) at Week 6
Description: Clinical Global Impressions - Severity: Bipolar Version (CGI-BP-S) score (depression) is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
Time Frame: 6 Weeks
Population: ITT population, excluding subjects from Japan Region
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-4199 200 mg | SEP-4199 400 mg | Placebo
Number analyzed (Participants) | 96 | 97 | 96
units on a scale | -2.020 (0.144) | -1.958 (0.138) | -1.739 (0.144)
Statistical Analysis 1: Comparison: SEP-4199 200 mg vs Placebo; Test type: Superiority; p = 0.143, Mixed Models Analysis — nominal p-value; Mean Difference (Final Values) = -0.281, 95% CI 2-sided [-0.658 to 0.095], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: SEP-4199 400 mg vs Placebo; Test type: Superiority; p = 0.243, Mixed Models Analysis — nominal p-value; Mean Difference (Final Values) = -0.219, 95% CI 2-sided [-0.588 to 0.150], Standard Error of Mean 0.187

ADVERSE EVENTS:
Time Frame: Up to 7 weeks
Description: Adverse events were untoward medical occurrences that occurred on or after the first dose of study medication.
Arm/Group | SEP-4199 200 mg | SEP-4199 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/114 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/113 | 0/114 | 1/114
Other Adverse Events (participants affected / at risk) | 21/113 | 23/114 | 29/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-4199 200 mg (N=113) | SEP-4199 400 mg (N=114) | Placebo (N=114)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-4199 200 mg (N=113) | SEP-4199 400 mg (N=114) | Placebo (N=114)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 6 (6)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 9 (9) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 3 (3) | 13 (16)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (5) | 7 (7)
Insomnia (Psychiatric disorders) | 5 (6) | 5 (6) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03543410/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT03543410/SAP_001.pdf